CLINICAL TRIAL: NCT07125794
Title: The Original Denis Brawn Brace Versus Its Modification for Management of Relapsed Idiopathic Clubfoot Following Ponseti Casting: A Retrospective Study.
Brief Title: Original Denis Brawn Brace Versus Its Modification for Management of Relapsed Idiopathic Clubfoot Following Ponseti Casting
Status: Recruiting | Type: Observational
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Mahmoud Mohamed Abdallah, Orthopedic Surgery, The General Authority for Teaching Hospitals and Institutes
Other Study IDs: HAH00072
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Denis Brawn Brace; Modification; Management; Idiopathic Clubfoot; Ponseti Casting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients who were managed with the original Denis Browne splint.
  Interventions: Procedure: Original Denis Browne splint
- Group II: Patients who were managed with the modified Denis Browne splint.
  Interventions: Procedure: Modified Denis Browne splint

INTERVENTIONS:
Procedure: Original Denis Browne splint — Patients who were managed with the original Denis Browne splint.
  Groups: Group I
Procedure: Modified Denis Browne splint — Patients who were managed with the modified Denis Browne splint.
  Groups: Group II

SUMMARY:
This study aims to compare the effectiveness of the original Denis Brawn brace to its modification in managing relapsed idiopathic clubfoot in patients following Ponseti casting.

DETAILED DESCRIPTION:
Clubfoot is an intricate deformity of the ankle and foot involving bony malalignment, adduction of the forefoot, and hindfoot varus, cavus, and equinus caused by contracture of soft tissues.

Lack of compliance causes the majority of relapse, as the child may have problems sleeping and wearing the Dennis Brown Splint; that is why parental counseling is vital and very much important in this regard.

Bracing plays a vital role in the maintenance of corrected club foot and allows the foot to achieve normal position after tenotomy, followed by serial casting. Bracing holds the foot not in a corrected but in an overcorrected position so that the normal position of the foot could be achieved after the correction. Without bracing, it is almost impossible for the physician or the surgeon to maintain the correction.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 to 5 years.
* Both sexes.
* Relapsed cases.
* Patients with idiopathic clubfoot.

Exclusion Criteria:

* Neurological or syndromic involvement.
* Presenting with skin or soft-tissue lesions around the foot and ankle.
* Inadequate documentation.
* Soft-tissue surgery is needed (except tendo-achilles tenotomy).
* Irregular plaster casting schedule.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This retrospective study will be carried out on 60 patients with idiopathic clubfoot after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Parents' compliance | 12 months post-procedure
  Parents' compliance will be classified into three grades as follows:
  * Grade 0: poor follow-up with a lack of commitment in bracing hours (bad compliance).
  * Grade 1: an intermittent follow-up with a good commitment in bracing hours (intermediate compliance).
  * Grade 2: a good follow-up with a strict commitment in bracing hours (good compliance).

SECONDARY OUTCOMES:
Efficacy in maintaining correction measured by the Pirani score | 12 months post-procedure
  The Pirani scoring system is reliable, quick, and easy to use, and provides a good forecast about the likely treatment for an individual foot. It involves evaluating six clinical signs of contracture, with scores ranging from 0 to 1 for each sign, and a higher score indicating a more severe deformity.
  All the patients treated will undergo thorough evaluation to find out other systemic diseases, and grading of the feet as per the modified Pirani scoring system.
Incidence of complications | 12 months post-procedure
  Incidence of complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.